CLINICAL TRIAL: NCT06795165
Title: A Single-center, Investigator-masked, Randomized, Placebo-controlled, Investigator-initiated Study of the Safety and Efficacy of Moxidectin Tablets for the Reduction of Demodex Eyelash Infestation.
Brief Title: Study of the Safety and Efficacy of Moxidectin Tablets for the Reduction of Demodex Eyelash Infestation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eye Research Foundation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MOX-001
Record Dates: First submitted 2025-01-22; First posted 2025-01-27 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Blepharitis
Keywords: blepharitis; demodex
MeSH Terms: conditions — Blepharitis | interventions — moxidectin; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Active (Active Comparator)
  Interventions: Drug: Moxidectin 2 MG Oral Tablet
- Active and Placebo (Experimental)
  Interventions: Drug: Moxidectin 2 MG Oral Tablet; Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Moxidectin 2 MG Oral Tablet — active medication
  Arms: Active; Active and Placebo
Drug: Placebo — placebo pills
  Arms: Active and Placebo; Placebo

SUMMARY:
A Single-Center, Investigator-Masked, Randomized, Placebo-Controlled, Investigator Initiated Study of the Safety and Efficacy of Moxidectin Tablets for the Reduction of Demodex Eyelash Infestation

ELIGIBILITY:
Inclusion Criteria:

- Active blepharitis with collarettes

Exclusion Criteria:

* Other clinically significant eye disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-02-02 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Collarette count | 6 weels
  Collarette Count

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Research Foundation, Inc., Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No